CLINICAL TRIAL: NCT00592709
Title: Analysis of Brain Tumors Using Matrix Assisted Laser Desorption/Ionization Mass Spectrometry
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Reid Thompson, Professor of Neurological Surgery, Vanderbilt University Medical Center
Other Study IDs: 030258
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Brain Diseases
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Brain Tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
We are collecting brain tissue specimens and blood samples from patients at Vanderbilt University Medical Center who are undergoing intracranial surgery to remove brain tissue, including brain tumors, tissue from epilepsy surgery and brain tissue removed during surgery for other non-cancerous types of brain tissus. These specimens will then be studied using a novel microscopic laser-directed protein mass spectrometric analysis, looking for unique protein signatures.

DETAILED DESCRIPTION:
We are collecting brain tissue specimens and blood samples from patients at Vanderbilt University Medical Center who are undergoing intracranial surgery to remove brain tissue, including brain tumors, tissue from epilepsy surgery and brain tissue removed during surgery for other non-cancerous types of brain tissus. These specimens will then be studied using a novel microscopic laser-directed protein mass spectrometric analysis. Data from different brain tissues including tumors of different histological sub-types will be analyzed for unique protein signatures. These protein signatures will then be statistically correlated with clinical data including time to tumor progression and response to therapy.

The goal of this study is to determine molecular patterns that will be more predictive of tumor behavior, thus leading to an improved understanding of the basic biology of these poorly understood cancers. This in turn, may lead to more refined therapies and improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of brain tumor or other non-cancerous tissue and are considered candidates fro a surgical procedure to biopsy or remove the brain tumor or other tissue type at Vanderbilt University Medical Center.
* Age 2 to 85

Exclusion Criteria:

* Patient or guardian that is unable to understand the informed consent process.

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Age 2 years through Age 85 years old
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2003-05; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measurement of proteomic signatures in brain tumor samples | immediately upon analysis of the sample
  measurement of proteomic signatures in brain tumor samples for unique protein signatures

CONTACTS AND LOCATIONS:
Overall Officials: Reid C. Thompson, MD, Principal Investigator — Vanderbilt University Medical Center, Department of Neurological Surgery
Locations (1):
- Vanderbilt University Medical Center, Department of Neurological Surgery, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No